CLINICAL TRIAL: NCT04189016
Title: Nasal Muco-ciliary Clearance Study With and Without Salt Inhalation Via a Salt Particle Inhaler at COPD, Asthma and Healthy Individuals
Brief Title: Nasal Muco-ciliary Clearance Study With and Without Salt Inhalation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liita Care ApS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: LC.002
Record Dates: First submitted 2019-11-28; First posted 2019-12-06 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Obstructive Airway Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salt particle inhaler with content (Active Comparator): Participants inhaling from a salt particle inhaler with content
  Interventions: Device: Inhalation from a salt particle inhaler with or without content
- Salt particle inhaler without content (Placebo Comparator): Participants inhaling from a salt particle inhaler without content
  Interventions: Device: Inhalation from a salt particle inhaler with or without content

INTERVENTIONS:
Device: Inhalation from a salt particle inhaler with or without content — Inhalation from inhaler with (active) or without (placebo) content

SUMMARY:
Investigating nasal muco-ciliary clearance by scintigraphy

DETAILED DESCRIPTION:
The velocity and the retention of the nasal muco-ciliary clearance is going to be investigated with a salt particle inhaler and a placebo by the method nasal scintigraphy.

The hypotheses is that nasal inhalation of salt particles enhance the nasal mucociliary clearance.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients (all severities in chronic, stable condition)
* Asthma patients (in stable condition without acute asthma symptoms)
* Healthy subjects, incl. smokers (no chronic nasal, upper or lower respiratory diseases)

Exclusion Criteria:

* Age under 18 years
* Upper respiratory tract infection / cold within the last 3 weeks and at least 3 weeks must pass from the person has become well to the examination
* Allergic / non-allergic rhinitis (hay fever)
* Chronic sinusitis
* Acute respiratory tract infection in antibiotic therapy
* Applied salt inhalation within the past month
* Pregnant or breastfeeding women
* Nuclear medical examination within the past month
* Cannot taste saccharin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Nasal Mucociliary Clearance | At study day 1 and 2
  Change in nasal mucociliary clearance velocity (mm/min) from placebo to salt inhalation
Nasal Mucociliary Clearance | At study day 1 and 2
  Change in nasal mucociliary clearance retention (%) from placebo to salt inhalation

SECONDARY OUTCOMES:
Spirometry | At the beginning and the end of study day 1 and 2
  Change in FEV! from placebo to saltinhalation
Saccharin test | At study day 1 and 2
  Change in time for saccharin transport

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Clin nuclear and physiolog dept., Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No